CLINICAL TRIAL: NCT00127959
Title: Virological and Clinical Anti-HBV Efficacy of Tenofovir and Emtricitabine in Antiretroviral Naïve Patients With HIV/HBV co-Infection
Brief Title: Virological and Clinical Anti-Hepatitis B Virus (HBV) Efficacy of Tenofovir and Emtricitabine in Patients With HIV/HBV co-Infection
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Antiviral Therapy Evaluation Center (Other)
Collaborators: Gilead Sciences (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IAT-0038-04
Record Dates: First submitted 2005-08-08; First posted 2005-08-09 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: HIV Infections; Hepatitis B
Keywords: HIV-1; HBV; treatment; tenofovir; emtricitabine; Treatment Naive; HIV-1 infection; Hepatitis B virus infection
MeSH Terms: conditions — HIV Infections; Hepatitis B | interventions — Tenofovir; Emtricitabine; Zidovudine; efavirenz

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: tenofovir
Drug: emtricitabine
Drug: zidovudine
Drug: efavirenz

SUMMARY:
This is a randomized multicentre trial of emtricitabine (FTC) versus tenofovir (TDF)/FTC in antiretroviral naive subjects with HIV/HBV co-infection over 48 weeks (Clinical Trial A).

Plus, a 12 week viral kinetic substudy comparing a subgroup of patients on Clinical Trial A is being conducted. (Substudy A1)

DETAILED DESCRIPTION:
This is a randomized multicentre trial of FTC vs TDF/FTC in antiretroviral naive subjects with HIV/HBV co-infection over 48 weeks (Clinical Trial A).

Plus, a 12 week viral kinetic substudy comparing a subgroup of patients on Clinical Trial A is being conducted. (Substudy A1)

Primary Objectives:

* To compare the proportion of subjects with HBV DNA levels below the limit of detection (<400 copies/ml) by week 48 in each treatment group

Secondary Objectives:

* To evaluate the emergence of HBV resistance at 48 weeks
* To compare the proportion of patients with undetectable HBV DNA at weeks 12 and 24 in each treatment group
* To compare the proportion of patients who achieve HBeAg and HBsAg seroconversion at weeks 12, 24 and 48 during the study
* To compare changes in ALT from baseline and the rate of hepatic cytolysis (ALT>5x ULN)
* To compare suppression of HIV-1 RNA and changes in CD4/CD8 counts over 48 weeks
* To compare the effect of therapy on histological changes in the liver and the presence of ccc-DNA

Enrollment:

* 24 patients in Clinical trial A (of whom 16 enter substudy A1).

Clinical Trial A:

* Patients with HIV/HBV co-infection who are naive to HIV/HBV therapy, have detectable HBV viraemia and are willing to start antiretroviral therapy.

Inclusion Criteria:

* Written informed consent
* Documented HIV infection
* Age 18 - 70 years
* HBV DNA > 106 copies/ml

Randomization:

* Arm 1: Zidovudine (AZT), emtricitabine (FTC), efavirenz (EFV)
* Arm 2: Tenofovir (TDF), emtricitabine (FTC), efavirenz (EFV)

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Documented HIV infection
* Age 18 - 70 years
* HBV DNA > 10E6 copies/ml
* ALT < 10 x ULN (upper limit of normal)
* Creatinine <= 2.0mg/dl
* Platelet count >= 50,000/mm3
* HIV-1 therapy naive
* No prior exposure to anti-HBV agents

Exclusion Criteria:

* Hepatitis C viral RNA (CV-RNA) positive or Anti-hepatitis A virus immunoglobulin M (HAV IgM) positive
* Acute hepatitis (serum ALT > 1000 U/L)
* Prior LAM, TDF, or adefovir dipivoxil (ADV) therapy
* Active opportunistic infection
* Pregnancy or lactation
* Other chronic liver disease
* Concurrent malignancy requiring cytotoxic chemotherapy
* Decompensated or Child's C cirrhosis
* Alfa-fetoprotein (AFP) > 3X ULN (unless negative computed tomography [CT] scan or magnetic resonance imaging [MRI] within 3 months of entry date)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2004-03; Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
HBV DNA suppression as measured by comparison of area under the curve (AUC) measurements after 48 weeks therapy

SECONDARY OUTCOMES:
Proportion of patients with undetectable HBV DNA in serum
Rate of hepatitis B e antigen (HBeAg) and hepatitis B surface antigen (HBsAg) seroconversion
Rate of emergence of lamivudine (LAM)-resistant HBV genotypes
Suppression of plasma HIV-RNA (< 50 copies/ml)
Changes in CD4+ /CD8+ cell counts
Presence of covalently closed circle DNA (cccDNA) on liver biopsy

CONTACTS AND LOCATIONS:
Overall Officials: Joep M.A. Lange, MD PhD, Study Chair — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA); Kiat Ruxrungtham, MD PhD, Principal Investigator — HIVNAT Bangkok; Jan Prins, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands